CLINICAL TRIAL: NCT04118686
Title: New Approaches for the Treatment of Early Stages of Cognitive Impairment in Neurodegenerative Diseases
Brief Title: Non-Pharmacological Treatments and Cognitive Impairment (NPT-CI2019)
Acronym: NPT-CI2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NPT-CI2019
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Cognitive Impairment
Keywords: Neurodegenerative disease; Cognitive decline; Non-pharmacological treatments; Cognitive training; Non-invasive brain stimulation
MeSH Terms: conditions — Cognitive Dysfunction; Neurodegenerative Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: A prospective, double-blind, randomized, parallel, controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The group receives CoRe software training plus non-invasive brain stimulation techniques (anodical tDCS / rTMS)
  Interventions: Other: CoRe software training plus non-invasive brain stimulation techniques (anodical tDCS / rTMS)
- Control group (Sham Comparator): The group receives CoRe software training plus sham non-invasive brain stimulation (sham tDCS/ sham rTMS)
  Interventions: Other: CoRe software training plus sham non-invasive brain stimulation (sham tDCS/ sham rTMS)

INTERVENTIONS:
Other: CoRe software training plus non-invasive brain stimulation techniques (anodical tDCS / rTMS) — CT program with Computerized cognitive training (CoRe) plus stimulation that modulates cortical activities by delivering strong magnetic pulses to the cortex through the scalp (rTMS) and weak electrical currents to the scalp to modulate neuronal transmembrane potential towards hyperpolarization or depolarization (tDCS).
  Arms: Experimental group
Other: CoRe software training plus sham non-invasive brain stimulation (sham tDCS/ sham rTMS) — CT program with Computerized cognitive training (CoRe) plus sham stimulation
  Arms: Control group

SUMMARY:
The prevalence of neurodegenerative diseases is expected to increase over the next years, in parallel with the aging of the world population. Therefore, it is important to identify new methods to prevent, delay or stop the neurodegenerative waterfall responsible for dementia conversion. To date, there is no fully proven pharmacological treatment for cognitive impairment and the available pharmacological armamentariums have limited efficacy because consist in symptomatic drugs with adverse side effects. On this point, non-pharmacological intervention may represent adjunctive therapy to medications in order to prevent or delay the onset of the cognitive deficits or dementia. This study aims to evaluate the effectiveness of a combined treatment protocol associating a Computerized cognitive training (CoRe) with non-invasive brain stimulation techniques: the transcranial Direct Current Stimulation (tDCS) or the repetitive Transcranial Magnetic Stimulation (rTMS). Patients with mild dementia or Mild Cognitive Impairment (MCI) are enrolled and randomly assigned to the experimental group (CoRe + anodic tDCS/rTMS) or control group (CoRe + sham tDCS/ sham rTMS). All patients are evaluated before (T0) and after (T1) treatment with an exhaustive neuropsychological assessment. Furthermore, follow-up visits are scheduled 6 months (T2) and 12 months (T3) after the end of the treatment.

DETAILED DESCRIPTION:
Non-pharmacological intervention may represent adjunctive therapy to medications in order to delay the onset of the cognitive deficits or dementia. Moreover, increasing evidence suggests that environmental and lifestyle factors (education, cognitive engagement, experience..) impact on cognitive functions and brain plasticity during the lifetime and also during aging. These modifiable factors moderate differences in cognitive aging and are protective for the development of dementia.

Among non-pharmacological approaches, previous studies observed a positive effect of Cognitive Training (CT) both in healthy elderly people and patients in the early stage of neurodegenerative diseases. Moreover, the advances in the development of Information & Communication Technologies has prompted the possibility to develop computer-based solution for the training of cognitive functions, being able to overcome traditional-training advantages. However, some issue remain unresolved and larger randomized controlled trials are necessary to examine long-term CT effects, due to the lack of longitudinal studies. Our previous data demonstrated that CT program with Computerized cognitive training (CoRe) software is safe and effective on cognition in patient with Parkinson Disease-Mild Cognitive Impairment, in the attempt of briefly stabilizing cognitive decline, delaying the downward trajectory.

Recently, different forms of non-invasive brain stimulation techniques have been applied to healthy older adults and patients with Alzheimer Disease (AD) in order to improve physiological and pathological aging-related cognitive impairments. Two main forms of non-invasive brain stimulation techniques are repetitive Transcranial Magnetic Stimulation (rTMS) and Transcranial Direct Current Stimulation (tDCS). rTMS is a painless, non-invasive method that modulates cortical activities by delivering strong magnetic pulses to the cortex through the scalp. Depending on stimulation parameters (e.g., duration, stimulus intensity, frequency), rTMS can enhance or suppress cortical excitability in targeted cortical regions. In general, high frequency rTMS facilitates cortical excitability whereas low frequency rTMS suppresses cortical excitability. tDCS delivers weak electrical currents to the scalp to modulate neuronal transmembrane potential towards hyperpolarization or depolarization, thereby altering plasticity in the stimulated brain regions. Depending on whether anodal or cathodal stimulation is applied, tDCS increases or decreases cortical excitability, respectively.These non-invasive brain stimulation techniques can be used alone or in combination with cognitive intervention programs. Some studies suggested that these non-invasive neurostimulation are able to enhance the effect of CT; however other studies yielded conflicting results, likely due to differences in stimulation parameters, experimental design and outcome measures. Thus, the overall efficacy of non-invasive neural stimulation as a therapeutic is still under debate.

In this frame, the primary goal of this double-blind randomized controlled trial is to assess whether the application of non-invasive brain stimulation techniques (tDCS or TMS) during the course of a computerized CT (on-line neurostimulation) enhances the effect on CT. Moreover, the follow-up visits allow to detect if the improvement are maintained over time and if this combined intervention affect the evolution of cognitive decline.

The treatment protocol consists of 12 sessions (4 session/week, 45 minutes/day) of CT with CoRe software (training memory and logical-executive functions) combined with on-line tDCS (anodic tDCS, 2mA for 20 minutes, versus sham tDCS applied to the cortical prefrontal cortex - DLPFC ) or rTMS (rTMS 20 Hz for 20 minutes versus sham TMS applied to DLPFC).

Patient with mild dementia or MCI are recruited from Neuropsychology/Alzheimer's Disease Assessment Unit and Neurorehabilitation Unit of IRCCS Mondino Foundation. The diagnosis of mild dementia or MCI is formulated on the basis of a comprehensive neuropsychological evaluation (baseline cognitive assessment - T0) according to the guidelines presented in the literature. The following standardized tests assessing different domains are used:

* global cognitive function: Mini-Mental State Examination (MMSE) and Montreal Montreal Overall Cognitive Assessment (MoCA);
* memory: verbal (Verbal Span; Digit Span) and spatial (Corsi's blocktapping test - CBTT) span; verbal long-term memory (Logical Memory Test immediate and delayed recall; Rey's 15-word test immediate and delayed recall); spatial long-term memory (Rey Complex Figure delayed recall - RCF-dr);
* logical-executive functions: non-verbal reasoning (Raven's Matrices 1947 - RM47); frontal functionality (Frontal Assessment Battery - FAB); semantic fluency (animals, fruits, car brands), phonological fluency (FAS);
* attention: visual selective attention (Attentive Matrices); simple speed processing and complex attention (Trail Making Test parts A - TMT A and part B - TMT B);
* visuospatial abilities: constructive apraxia Rey Complex Figure copy - RCF-copy.

The same battery is also used at follow-up visits; parallel versions are applied when available (verbal long-term memory tests), in order to avoid the learning effect. All the test scores are corrected for age, sex, and education and compared with the values available for the Italian population.

At the baseline, the cognitive reserve is assessed using Cognitive Reserve Index questionnaire (CRIq). The patients' functional status is assessed using Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) at the baseline and at the last follow-up visit after one year (T3). Moreover, mood is assessed using the Beck Depression Inventory (BDI) at the baseline and at the follow-up visits (T1, T2 and T3), while quality of life were assessed using the 36-Item Short Form Health Survey questionnaire (SF-36) at the baseline and at the follow-up visits six months (T2) and one year (T3) after training.

All the patients recruited undergo baseline cognitive assessment (T0). Patients who met the inclusion and exclusion criteria are enrolled and randomly assigned to the experimental group (CoRE + anodic tDCS/rTMS) or control group (CoRe + sham tDCS/rTMS).

ELIGIBILITY:
Inclusion Criteria:

* presence of mild dementia or mild cognitive impairment;
* age between 50 and 85 years;
* educational level ≥ 5 years.

Exclusion Criteria:

* pre-existing cognitive impairment (e.g. aphasia, neglect);
* severe disturbances in consciousness;
* concomitant severe psychiatric disease or others neurological conditions (e.g. depression and behavioural disorders).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive functioning measured by Mini-Mental State Examination (MMSE) | After 3 -week intervention program (T1), 6 months (T2) and 1 year (T3) after the end of intervention program
  It is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. The score is between 0-30. Lower score is worse cognitive functioning.
Change in global cognitive functioning measured by Montreal Overall Cognitive Assessment (MoCA) | After 3 -week intervention program (T1), 6 months (T2) and 1 year (T3) after the end of intervention program
  It is a widely used screening assessment for detecting cognitive impairment. It assesses several cognitive domains:
  The short-term memory recall task (5 points). Visuospatial abilities a clock-drawing task (3 points) and a three-dimensional cube copy (1 point). Multiple aspects of executive functions are assessed using an alternation task adapted from the trail-making B task (1 point), a phonemic fluency task (1 point), and a two-item verbal abstraction task (2 points). Attention, concentration, and working memory are evaluated using a three-item confrontation naming task with low-familiarity animals (3 points), repetition of two syntactically complex sentences (2 points), and the aforementioned fluency task. Finally, orientation to time and place (6 points). Low score is worse outcome.

SECONDARY OUTCOMES:
Change in memory | After 3 -week intervention program (T1), 6 months (T2) and 1 year (T3) after the end of intervention program
  Verbal and spatial span; verbal long-ter memory; spatial long-term memory by using scales. Higher scores are better outcomes.
Change in executive functions | After 3 -week intervention program (T1), 6 months (T2) and 1 year (T3) after the end of intervention program
  Logical-executive functions; attention; visuospatial abilities by using scale. Higher scorea are better outcomes.
Change in mood (assessed by Beck Depression Inventory - BDI) | After 3 -week intervention program (T1), 6 months (T2) and 1 year (T3) after the end of intervention program
  Contains 21 questions. The items are rated on a 4-point severity scale (0-3) and are summed to give a total score (range 0-63). A higher score denotes more severe depression.
Change in Quality of Life (assessed by Short Form-36 Health Survey - SF - 36) | After 3 -week intervention program (T1), 6 months (T2) and 1 year (T3) after the end of intervention program
  Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carriers equal weight. Low score is worse quality of life.
Change in the evolution of cognitive profile (assessed by Clinical Dementia Rating Scale - CDR) | After 3 -week intervention program (T1), 6 months (T2) and 1 year (T3) after the end of intervention program
  CDR is a widely utilized clinical tool for grading the relative severity of dementia with scores that range from 0 (no impairment) to 3 (severe impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sinforiani, MD, Principal Investigator — Struttura Semplice Neuropsicologia Clinica/Centro UVA
Locations (1):
- Struttura Semplice Neuropsicologia Clinica/ Centro UVA, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Background] Coyle H, Traynor V, Solowij N. Computerized and virtual reality cognitive training for individuals at high risk of cognitive decline: systematic review of the literature. Am J Geriatr Psychiatry. 2015 Apr;23(4):335-359. doi: 10.1016/j.jagp.2014.04.009. Epub 2014 May 14. PMID 24998488
- [Background] Bernini S, Alloni A, Panzarasa S, Picascia M, Quaglini S, Tassorelli C, Sinforiani E. A computer-based cognitive training in Mild Cognitive Impairment in Parkinson's Disease. NeuroRehabilitation. 2019;44(4):555-567. doi: 10.3233/NRE-192714. PMID 31256092
- [Background] Prehn K, Floel A. Potentials and limits to enhance cognitive functions in healthy and pathological aging by tDCS. Front Cell Neurosci. 2015 Sep 14;9:355. doi: 10.3389/fncel.2015.00355. eCollection 2015. PMID 26441526
- [Background] Hsu WY, Ku Y, Zanto TP, Gazzaley A. Effects of noninvasive brain stimulation on cognitive function in healthy aging and Alzheimer's disease: a systematic review and meta-analysis. Neurobiol Aging. 2015 Aug;36(8):2348-59. doi: 10.1016/j.neurobiolaging.2015.04.016. Epub 2015 May 1. PMID 26022770
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Litvan I, Goldman JG, Troster AI, Schmand BA, Weintraub D, Petersen RC, Mollenhauer B, Adler CH, Marder K, Williams-Gray CH, Aarsland D, Kulisevsky J, Rodriguez-Oroz MC, Burn DJ, Barker RA, Emre M. Diagnostic criteria for mild cognitive impairment in Parkinson's disease: Movement Disorder Society Task Force guidelines. Mov Disord. 2012 Mar;27(3):349-56. doi: 10.1002/mds.24893. Epub 2012 Jan 24. PMID 22275317
- [Derived] Rodella C, Bernini S, Panzarasa S, Sinforiani E, Picascia M, Quaglini S, Cavallini E, Vecchi T, Tassorelli C, Bottiroli S. A double-blind randomized controlled trial combining cognitive training (CoRe) and neurostimulation (tDCS) in the early stages of cognitive impairment. Aging Clin Exp Res. 2022 Jan;34(1):73-83. doi: 10.1007/s40520-021-01912-0. Epub 2021 Jun 22. PMID 34156651